CLINICAL TRIAL: NCT03656029
Title: Dose-dependent Effects of Smoked Cannabis on Simulated Driving Performance
Brief Title: Dose-response of Cannabis and Driving
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 007-2018
Record Dates: First submitted 2018-08-08; First posted 2018-09-04 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Driving Impaired; Cognitive Impairment; Abuse Cannabis
MeSH Terms: conditions — Cognitive Dysfunction; Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: This will be a within-subjects, counterbalanced, placebo-controlled study of placebo or 3 doses of cannabis
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Placebo (Placebo Comparator): Participants will smoke a single smoked placebo (<0.1% THC) cannabis cigarette
  Interventions: Drug: Placebo
- low dose (Active Comparator): Participants will smoke a single low dose (6.25% THC) of smoked cannabis cigarette
  Interventions: Drug: Cannabis
- middle dose (Active Comparator): Participants will smoke a single intermediate dose (12.5% THC) of smoked cannabis cigarette
  Interventions: Drug: Cannabis
- high dose (Active Comparator): Participants will smoke a single high dose (22% THC) of smoked cannabis cigarette
  Interventions: Drug: Cannabis

INTERVENTIONS:
Drug: Cannabis — Participants will smoke as much of the cigarette as they wish
  Arms: high dose; low dose; middle dose
Drug: Placebo — Participants will smoke a placebo cigarette
  Arms: Placebo

SUMMARY:
Epidemiological studies have established a link between collisions while driving and cannabis use. With the changing legal landscape around cannabis, there is much interest in determining per se limits of cannabis while driving. The present study will evaluate driving on a driving simulator after smoking placebo or cannabis with 3 different levels of THC. THC is the active component in cannabis and blood, urine and oral fluid levels of THC will be correlated with driving impairment.

DETAILED DESCRIPTION:
Participants will attend the laboratory for 4 separate sessions, separated by about a week. In each session, participants will receive one of 3 doses of smoked cannabis or a placebo. Participants will not know which dose they are receiving. Participants will complete questionnaires, do cognitive tests and drive on a driving simulator before and after smoking the cannabis or placebo cigarette. Blood, urine and oral fluid will be collected throughout the 7-8 hour session to determine levels of THC and its metabolites. These values will be correlated with measures of driving impairment.

ELIGIBILITY:
Inclusion Criteria:

* Near daily use of cannabis (1-5 days/week) confirmed by self-report and urine screening
* Has held a class G2 or G licence (or equivalent from another jurisdiction) for at least 12 months
* Willing to abstain from using cannabis for 72 hours prior to each practice or test session
* Willing to abstain from alcohol for 48 hours prior to each session, and to abstain from all other drugs not medically required for the duration of the study (beginning 48 hours prior to the practice session)
* Provides written and informed consent

Exclusion Criteria:

* Diagnosis of severe medical or psychiatric condition
* Meets criteria for current or lifetime alcohol or other substance use disorder, except tobacco use disorder and caffeine use disorder
* Regular user of medication that may affect cognitive functioning and/or driver performance
* Family history of schizophrenia or other psychotic disorder
* Pregnant, looking to become pregnant, or breastfeeding

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Mean speed | Change in speed of driving between the time before smoking the cigarette and either 30 or 90 minutes after smoking the cigarette
  Speed of driving the simulator

SECONDARY OUTCOMES:
Standard deviation of lateral position | Change in measure from before smoking the cigarette to either 30 or 90 minutes after smoking
  Driving measures
reaction time | Change in measure from before smoking the cigarette to either 30 or 90 minutes after smoking
  Driving measures
Blood concentrations of THC and metabolites | Change from before smoking cigarette to various time points after smoking: 5 minutes, 15 minutes, 30 minutes, 60 minutes, 90 minutes, 2hours, 3 hours, 4 hours, 5 hours and 6 hours
  Blood will be taken to determine how much THC entered the blood
Oral fluid concentrations of THC and metabolites | Change from levels before smoking to 4 time points after smoking: 30 minutes, 90 minutes, 2 hours and 6 hours
  Participants will provide oral fluid to determine how much THC is in the oral fluid
Systolic and Diastolic Blood pressure | Change from before smoking to a number of time points after smoking: 5 minutes, 15 minutes, 30 minutes, 60 minutes, 90 minutes, 2hours, 3 hours, 4 hours, 5 hours and 6 hours
  Vital signs
Heart rate | Change from before smoking to a number of time points after smoking: 5 minutes, 15 minutes, 30 minutes, 60 minutes, 90 minutes, 2hours, 3 hours, 4 hours, 5 hours and 6 hours
  Vital signs
Respirations | Change from before smoking to a number of time points after smoking: 5 minutes, 15 minutes, 30 minutes, 60 minutes, 90 minutes, 2hours, 3 hours, 4 hours, 5 hours and 6 hours
  Vital signs
Temperature | Change from before smoking to a number of time points after smoking: 5 minutes, 15 minutes, 30 minutes, 60 minutes, 90 minutes, 2hours, 3 hours, 4 hours, 5 hours and 6 hours
  Vital signs
Visual Analog Scales | Change from before smoking to a number of time points after smoking: 5 minutes, 15 minutes, 30 minutes, 60 minutes, 90 minutes, 2hours, 3 hours, 4 hours, 5 hours and 6 hours
  Tests designed to assess the degree of subjective effects of the drug. The questions will be scored on a scale from 0 to 100 and will consist of: 'I like this drug effect', 'this feels like cannabis', 'I feel this effect', 'I feel this high', 'I feel the good effects', 'I feel the bad effects', 'I feel the rush'
Verbal free recall test | Change from pre-smoking levels to those observed 60 minutes after smoking
  Test of memory: Participants will be asked to recall words that are read from a list
Useful field of view | Change from pre-smoking levels to those observed 60 minutes after smoking
  A computer test for visual processing speed, selective and divided attention

CONTACTS AND LOCATIONS:
Overall Officials: Bruna Brands, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Center for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No